CLINICAL TRIAL: NCT01568385
Title: A Unblinded Study of TAK-438 (20 mg) for Prevention of Recurrence of Gastric or Duodenal Ulcer During Long-Term Non-Steroid Anti-Inflammatory Drug (NSAID) Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: TAK-438/OCT-303; U1111-1128-5905 (Registry Identifier: WHO); JapicCTI-121789 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-02

CONDITIONS: Gastric Ulcer; Duodenal Ulcer
Keywords: Gastric or duodenal ulcer
MeSH Terms: conditions — Stomach Ulcer; Duodenal Ulcer | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

ARMS (1):
- TAK-438 20 mg QD (Experimental)
  Interventions: Drug: TAK-438

INTERVENTIONS:
Drug: TAK-438

SUMMARY:
The purpose of this study is to study the safety and efficacy of TAK-438, once daily (QD), in participants with a history of gastric or duodenal ulcer requiring long-term NSAID therapy will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who, in the opinion of the principal investigator or subinvestigator, are capable of understanding the details of the study and complying with them.
2. Prior to study commencement, participants who are capable of signing and dating the information/consent form.
3. Participants with a chronic disease (rheumatoid arthritis, osteoarthritis, etc.) which requires continuous NSAID oral therapy for pain control during treatment period.
4. Participants who meet either 1 or 2 below according to gastric or duodenal endoscopy:

   * Ulcer scar (defined, in this study, as regenerative mucosa, convergence of mucosal fold, gastric wall transformation, etc) has been confirmed during endoscopy on the study drug initiation day (Visit 2).
   * Ulcer (mucosal defects of 3 mm or larger with white moss) or ulcer scar has been endoscopically confirmed before the study drug initiation day (Visit 2).
5. Outpatient participants (inpatients for examinations are acceptable)
6. Women with child-bearing potential must agree to routinely take appropriate contraceptive measures throughout treatment period, from giving consent to the study until 4 weeks after the final dose

Exclusion Criteria:

1. Participants who received treatment with another study drug (including approved drugs under post-marketing surveillance) within 84 days prior to commencement of screening
2. Participants who have previously received TAK-438 in a clinical study or as a treatment
3. Participants who are employees of institutions participating in this study and family members of such employees, participants in a dependent relationship with employees of institutions involved in conduct of the study (e.g., spouse, parent, child, sibling), and participants who are under duress in giving their consent
4. Participants who have donated 400 mL or more of blood within 90 days prior to the commencement of screening
5. Participants with a plan to change the type, dosage or administration of NSAID
6. Participants with ulcer (mucosal defects of 3 mm or larger with white moss) or active hemorrhage confirmed during gastric or duodenal endoscopy on the study drug initiation day (Visit 2)
7. Participants with small intestinal hemorrhage, large intestinal hemorrhage, or gastrointestinal hemorrhage of unknown cause
8. Participants with a history of surgery or scheduled surgery influencing gastric acid secretion (resection of upper gastrointestinal tract or vagotomy etc)
9. Participants with a history or complication of Zollinger-Ellison syndrome, or other gastric acid hypersecretion disorders
10. Participants with a history or complication of aspirin asthma
11. Participants who have a history of hypersensitivity or allergy to TAK-438 (including its excipients) or NSAIDs
12. Participants with current use of illicit drug or a history of drug abuse. and/or alcohol dependence within one year prior to the commencement of screening
13. Participants who require treatment with prohibited concomitant drugs or therapies (see 7.3)
14. Female participants who are pregnant or lactating; those who plan to become pregnant or donate ova during treatment period, from giving consent until 4 weeks after final dose
15. Participants with serious central nervous system disorders, cardiovascular disease, pulmonary disease, hepatic disease, renal disease, metabolic disease, gastrointestinal disorders, urinary disorders, endocrine disease, or blood dyscrasia
16. Participants who plan to undergo surgery requiring hospitalization or requires surgery during the study period.
17. Participants with a history of a malignancy (or treatment thereof) within 5 years prior to the commencement of screening; however, participants with completely cured basal cell carcinoma of skin or carcinoma in situ of the cervix may be included in the study.
18. Participants with acquired immune deficiency syndrome (AIDS; including HIV carriers) or hepatitis (including viral hepatitis carriers [HBs antigen or HCV antibody positive]); however, participants who are hepatitis C virus (HCV) antigen negative or HCV-RNA negative may be included in the study.
19. Participants who meet either of the following laboratory test values at the beginning of screening (Visit 1)

    * Serum creatinine value: higher than 2 mg/dL
    * Alanine transaminase (ALT) or aspartate aminotransferase (AST): higher than 2.5 × the upper limit of normal
    * Total bilirubin: higher than 2.0 × the upper limit of normal

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Adverse Event | 24 weeks

CONTACTS AND LOCATIONS:
Locations (18):
- Japan (18):
  - Funabashi-shi, Chiba
  - Noda, Chiba
  - Fukuoka, Fukuoka
  - Annaka-shi, Gunma
  - Hiroshima, Hiroshima
  - Hakodate-shi, Hokkaido
  - Kitahiroshima-shi, Hokkaido
  - Sapporo, Hokkaido
  - Yubari-gun, Hokkaido
  - Kanazawa, Ishikawa-ken
  - Sanuki-shi, Kagawa-ken
  - Yashiro-shi, Kumamoto
  - Nagasaki, Nagasaki
  - Sasebo-shi, Nagasaki
  - Fuchu-shi, Tokyo
  - Katsushika-ku, Tokyo
  - Meguro-ku, Tokyo
  - Nakano-ku, Tokyo